CLINICAL TRIAL: NCT06725823
Title: Therapeutic Effect of Shoulder Anterior Capsular Block (SHAC) Versus Suprascapular Nerve Block in Patients With Frozen Shoulder
Brief Title: Therapeutic Effect of Shoulder Anterior Capsular Block Versus Suprascapular Nerve Block in Patients With Frozen Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ayat Abdulwahab Othman, Assistant lecturer of Physical Medicine, Rheumatology &Rehabilitation, Sohag University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-24-11__2MD
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: The study will include 50 patients with frozen shoulder with no healthy volunteer, Patients in this study will be randomized into two groups according to the treatment performed Shoulder anterior capsular block group and Suprascapular nerve block group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: patients will not be aware about which type of intervention they will recieve also the care provider and outcome assessor will be not aware about type of intervention patients will recieve
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprascapular nerve block group (Active Comparator): Patients will be placed in lateral position by using A high - frequency linear ultrasound probe will be placed approximately 2 cm medial to the medial border of the acromion and about 2 cm cranial to the superior margin of the scapular spine the needle will be inserted .The tip of the needle will be placed at the floor of the supraspinatus fossa where the nerve has passed
  Interventions: Procedure: suprascapular nerve block group
- shoulder anterior capsular block group (Active Comparator): Ultrasound guided injection For the SHAC block, with the patient in a beach-chair position and with the arm in extension, the subscapularis muscle is stretched posteriorly and becomes easily visible. With external rotation and abduction, the coracobrachialis and the biceps brachii muscles are displaced, allowing the visualization of the interfascial space between the deep lamina of the deltoid muscle fascia and the superficial lamina of the subscapularis fascia.Once the injection into the fascial space is achieved, the investigators can proceed towards the glenohumeral pericapsular space by crossing the subscapularis muscle with the needle. By injecting the pericapsular space, the investigators reach the terminal articular branches indistinctly from their origin. Furthermore, through the Weitbrecht foramen, a natural capsular foramen between the upper and middle glenohumeral ligaments, we also reach the intra-articular space .
  Interventions: Procedure: shoulder anterior capsular block group

INTERVENTIONS:
Procedure: suprascapular nerve block group — A volume of (10 ml) of 2% lidocaine (7ml), 3% Mepivacaine (2ml), 1 ml methyl-prednisolone acetate (40 mg) will be injected to both groups.
  Arms: suprascapular nerve block group
Procedure: shoulder anterior capsular block group — A volume of (10ml) of 2% lidocaine (7ml), 3% Mepivacaine (2ml), 1 ml methyl-prednisolone acetate (40mg) will be injected to both groups.
  Arms: shoulder anterior capsular block group

SUMMARY:
he study will include 50 patients with frozen shoulder with no healthy volunteer , Patients in this study will be randomized into two groups suprascapular nerve block and Shoulder anterior capsular block

DETAILED DESCRIPTION:
The study will include 50 patients with frozen shoulder with no healthy volunteer , Patients in this study will be randomized into two groups according to the treatment performed .

Shoulder anterior capsular block group

Description:

Ultrasound guided injection For the SHAC block, with the patient in a beach-chair position and with the arm in extension, the subscapularis muscle is stretched posteriorly and becomes easily visible. With external rotation and abduction, the coracobrachialis and the biceps brachii muscles are displaced, allowing the visualization of the interfascial space between the deep lamina of the deltoid muscle fascia and the superficial lamina of the subscapularis fascia.Once the injection into the fascial space is achieved, the investigators can proceed towards the glenohumeral pericapsular space by crossing the subscapularis muscle with the needle. By injecting the pericapsular space, the investigators reach the terminal articular branches indistinctly from their origin. Furthermore, through the Weitbrecht foramen, a natural capsular foramen between the upper and middle glenohumeral ligaments, we also reach the intra-articular space .

Suprascapular nerve block group

Description:

Patients will be placed in lateral position by using A high - frequency linear ultrasound probe will be placed approximately 2 cm medial to the medial border of the acromion and about 2 cm cranial to the superior margin of the scapular spine the needle will be inserted .The tip of the needle will be placed at the floor of the supraspinatus fossa where the nerve has passed

* A volume of (10ml) of 2% lidocaine (2ml), 3% Mepivacaine (2ml) , 1 ml methyl-prednisolone acetate (40 mg) and dextrose 5% (5ml) will be injected to both groups.
* All patients in both groups will receive immediate stretching exercises and post injection 3 times weekly followed by home exercises

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.

  * Both sexes, males and females.
  * History of complaint >6 weeks
  * Restricted shoulder movement unilaterally in at least 2 planes including abduction, external rotation, and internal rotation and restricted passive movement.

Exclusion Criteria:

* Patient refusal.

  * -Allergy to local anaesthetics.
  * -Infection at the site of injection .
  * -Coagulopathy
  * -Prolonged opioid medication
  * -Pregnancy
  * -Acute trauma, fracture of the shoulder
  * People who had received an intra-articular shoulder injection within the last 6 months.
  * Patients with tendon tear

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain (Visual analogue scale) | at baseline and post-procedure at 1, 3 and 6 months.
  s a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
total pain scores | at baseline and post-procedure at 1, 3 and 6 months.
  is a combination of simple pain score, radiation, and sleep disturbance score
shoulder pain disability index | at baseline and post-procedure at 1, 3 and 6 months.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
active range of movement of the shoulder joint | at baseline and post-procedure at 1, 3 and 6 months.
  The active and passive range of abduction, adduction, flexion , extension , internal rotation and external rotation will be measured using goniometry

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Basta M, Sanganeria T, Varacallo MA. Anatomy, Shoulder and Upper Limb, Suprascapular Nerve. 2022 Oct 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557880/ PMID 32491803
- [Result] Brindisino F, Girardi G, Crestani M, Assenza R, Andriesse A, Giovannico G, Pellicciari L, Salomon M, Venturin D. Rehabilitation in subjects with frozen shoulder: a survey of current (2023) clinical practice of Italian physiotherapists. BMC Musculoskelet Disord. 2024 Jul 23;25(1):573. doi: 10.1186/s12891-024-07682-w. PMID 39044183
- [Result] Millar NL, Meakins A, Struyf F, Willmore E, Campbell AL, Kirwan PD, Akbar M, Moore L, Ronquillo JC, Murrell GAC, Rodeo SA. Frozen shoulder. Nat Rev Dis Primers. 2022 Sep 8;8(1):59. doi: 10.1038/s41572-022-00386-2. PMID 36075904